CLINICAL TRIAL: NCT00737685
Title: Fludarabine, Cyclophosphamide Plus Thymoglobulin Conditioning Regimen for Unrelated Bone Marrow (or Mobilized Peripheral Blood) Transplantation in Severe Aplastic Anemia
Brief Title: Flu+CPM+rATG Conditioning Regimes for Unrelated Bone Marrow Transplantation (UBMT)(or Mobilized Peripheral Blood)in Severe Aplastic Anemia (SAA)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The Korean Society of Pediatric Hematology Oncology (Network)
Responsible Party: Hyo Seop Ahn, Seoul Natioanl University Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KSPHO-SCT0401
Record Dates: First submitted 2008-08-18; First posted 2008-08-19 (Estimated); Last update posted 2012-03-26 (Estimated); Status verified 2012-03

CONDITIONS: Anemia, Aplastic
Keywords: Pediatric; UBMT; Severe
MeSH Terms: conditions — Anemia, Aplastic; Lymphoma, Follicular | interventions — Cyclophosphamide; fludarabine; thymoglobulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fludarabine (Experimental)
  Interventions: Drug: cyclophosphamide, fludarabine , thymoglobulin

INTERVENTIONS:
Drug: cyclophosphamide, fludarabine , thymoglobulin — cyclophosphamide (50 mg/kg once daily i.v. on days -9, -8, -7 & -6) fludarabine (30 mg/m2 once daily i.v. on days -5, -4, -3 & -2) thymoglobulin (2.5 mg/kg once daily i.v. on days -3, -2 & -1)

SUMMARY:
Anti-thymocyte globulin (ATG) has been used in severe aplastic anemia as a part of the conditioning regimen. Among the many kinds of ATG preparations, thymoglobulin had been found to be more effective in preventing GVHD and rejection of organ transplants. As the fludarabine based conditioning regimens without total body irradiation have been reported to be promising for BMT/PBSCT from alternative donors in SAA, thymoglobulin was added to fludarabine and cyclophosphamide conditioning to reduce GVHD and to allow good engraftment in UBMT/UPBSCT.

DETAILED DESCRIPTION:
GVHD prophylaxis recommendation tacrolimus (0.03 mg/kg/day i.v. by continuous infusion from day -2 and taper with an oral form until 1 year after BMT/PBSCT) methotrexate (15 mg/m2 i.v. on days 1 and 10 mg/m2 i.v. on days 3, 6, 11)

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of severe aplastic anemia defined by any two or three peripheral blood criteria
* and either marrow criterion.
* Peripheral blood

  1. Neutrophils < 0.5 x 109/l
  2. Platelets < 20 x 109/l
  3. Corrected reticulocytes < 1%
* Bone marrow

  1. Severe hypocellularity (< 25%)
  2. Moderate hypocellularity (25-30%) with hematopoietic cells representing < 30% of residual cells
* No prior hematopoietic stem cell transplantation.
* Age: no limits.
* Performance status: ECOG 0-2.
* Patients must be free of significant functional deficits in major organs, but the following eligibility criteria may be modified in individual cases.

  1. Heart: a shortening fraction > 30%, ejection fraction > 45%.
  2. Liver: total bilirubin < 2 × upper limit of normal; ALT < 3 × upper limit of normal.
  3. Kidney: creatinine <2 × normal or a creatinine clearance (GFR) > 60 ml/min/1.73m2.
* Patients must lack any active viral infections or active fungal infection.
* Appropriate donor is available: Matched in 6/6 of A, B, DR loci.
* Patients (or one of parents if patients age < 19) should sign informed consent.

Exclusion Criteria:

* Pregnant or nursing women.
* Malignant or nonmalignant illness that is uncontrolled or whose control may be jeopardized by complications of study therapy.
* Psychiatric disorder that would preclude compliance.
* Congenital aplastic anemia including Fanconi anemia.
* Manipulated bone marrow.

Max Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2006-01; Primary Completion 2012-08 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
To evaluate the engraftment potential, incidence and severity of acute graft versus host disease,toxicity of conditioning regimen for UBMT in SAA. | From Jan. 1. 2006 to Dec. 31. 2008. For 3 years.
To evaluate overall and EFS follow-up of 1 year after UBMT/PBSCT. | From Jan. 1. 2006 to Dec. 31. 2008. For 3 years

SECONDARY OUTCOMES:
To evaluate chronic GVHD and immunologic recovery after UBMT/PBSCT. and the efficacy of UBMT/PBSCT before immuno-suppressive therapy with anti-thymocyte globulin in severe aplastic anemia and long term toxicity of non-TBI based conditioning | From Jan. 1. 2006 to Dec. 31. 2008. For 3 years.

CONTACTS AND LOCATIONS:
Overall Officials: Hyo Seop Ahn, M.D, Ph.D, Principal Investigator — The Korean Society of Pediatric Hematology Oncology
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Kang HJ, Shin HY, Park JE, Chung NG, Cho B, Kim HK, Kim SY, Lee YH, Lim YT, Yoo KH, Sung KW, Koo HH, Im HJ, Seo JJ, Park SK, Ahn HS; Korean Society of Pediatric Hematology-Oncology. Successful engraftment with fludarabine, cyclophosphamide, and thymoglobulin conditioning regimen in unrelated transplantation for severe aplastic anemia: A phase II prospective multicenter study. Biol Blood Marrow Transplant. 2010 Nov;16(11):1582-8. doi: 10.1016/j.bbmt.2010.05.010. Epub 2010 May 26. PMID 20685256